CLINICAL TRIAL: NCT06606756
Title: CEDATA GPGE Patient Registry for Children and Adolescents with IBD
Brief Title: CEDATA GPGE - a Patient Registry for Children and Adolescents with Inflammatory Bowel Disease
Acronym: CEDATA GPGE
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Jan De Laffolie, Head Paed Gastroenterology, University of Giessen
Other Study IDs: CEDATA GPGE
Record Dates: First submitted 2024-09-04; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: paediatric; crohns disease; ulcerative colitis; quality improvement; patient registry
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: Patient Registry without intervention — This is a patient registry that collects real world data without intervening with therapeutic decision
Other: Digital Registry and Feedback on clinical data — The data is entered via a validated online platform and is provided back to the center in aggregated form

SUMMARY:
CEDATA GPGE collects clinical data of children and adolescents with IBD from paediatric gastroenterology centers in german-speaking countries.

Data is obtained from participating centers in pseudonymized way via an online platform at the beginning and during followup of the disease. The leading working group of the paediatric gastroenterology society GPGE e.V. includes 15 experts in the field who meet twice yearly and coordinate research and quality improvement initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory Bowel Disease

Exclusion Criteria:

* none

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and adolescents with IBD
Sampling Method: Non-Probability Sample
Enrollment: 6300 (Estimated)
Dates: Start 2004-09-01 (Actual); Primary Completion 2034-12-01 (Estimated); Study Completion 2034-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission | any
  Clinical Remission - absence of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University Giessen, Giessen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Laffolie J, Koletzko S, Buderus S, Classen M, Posovszky C, Rodeck B, Keller KM, Lang T, Hauer A; CEDATA GPGE Study Group. Lack of Correlation of Mean Corpuscular Volume to White Blood Cell Ratio to Thiopurine Levels. J Pediatr Gastroenterol Nutr. 2020 May;70(5):e107-e110. doi: 10.1097/MPG.0000000000002662. No abstract available. PMID 32079979
- [Background] Kern I, Schoffer O, Richter T, Kiess W, Flemming G, Winkler U, Quietzsch J, Wenzel O, Zurek M, Manuwald U, Hegewald J, Li S, Weidner J, de Laffolie J, Zimmer KP, Kugler J, Laass MW, Rothe U. Current and projected incidence trends of pediatric-onset inflammatory bowel disease in Germany based on the Saxon Pediatric IBD Registry 2000-2014 -a 15-year evaluation of trends. PLoS One. 2022 Sep 9;17(9):e0274117. doi: 10.1371/journal.pone.0274117. eCollection 2022. PMID 36084003
- [Background] Kern I, Schoffer O, Kiess W, Henker J, Laass MW, Winkler U, Quietzsch J, Wenzel O, Zurek M, Buttner K, Fischer P, de Laffolie J, Manuwald U, Stange T, Zenker R, Weidner J, Zimmer KP, Kunath H, Kugler J, Richter T, Rothe U. Incidence trends of pediatric onset inflammatory bowel disease in the years 2000-2009 in Saxony, Germany-first results of the Saxon Pediatric IBD Registry. PLoS One. 2021 Jan 4;16(1):e0243774. doi: 10.1371/journal.pone.0243774. eCollection 2021. PMID 33395450
- [Background] Schiller B, Wirthgen E, Weber F, Schiller S, Radke M, Classen M, Dabritz J; CEDATA-GPGE Study Group. Fecal calprotectin and platelet count predict histologic disease activity in pediatric ulcerative colitis: results from a projection-predictive feature selection. Eur J Pediatr. 2024 Aug;183(8):3277-3288. doi: 10.1007/s00431-024-05554-y. Epub 2024 May 6. PMID 38709314
- [Background] de Laffolie J, Zimmer KP, Sohrabi K, Hauer AC. Running Behind "POPO"-Impact of Predictors of Poor Outcome for Treatment Stratification in Pediatric Crohn's Disease. Front Med (Lausanne). 2021 Aug 27;8:644003. doi: 10.3389/fmed.2021.644003. eCollection 2021. PMID 34513855
- [Background] Tischler L, Boerkoel A, Krause H, van den Berg N, de Laffolie J. The Care of Children and Adolescents with Chronic Inflammatory Bowel Disease: A Cluster-Randomized Trial on Improving the Guideline Conformity of Treatment by the Use of the CEDATA-GPGE Patient Registry. Dtsch Arztebl Int. 2024 Sep 20;121(19):627-633. doi: 10.3238/arztebl.m2024.0168. PMID 39163213
- [Background] de Laffolie J, Laass MW, Scholz D, Zimmer KP, Buderus S; CEDATA-GPGE Study Group. Prevalence of Anemia in Pediatric IBD Patients and Impact on Disease Severity: Results of the Pediatric IBD-Registry CEDATA-GPGE(R). Gastroenterol Res Pract. 2017;2017:8424628. doi: 10.1155/2017/8424628. Epub 2017 Dec 5. PMID 29358946
- [Background] de Laffolie J, Schwerd T, Simon A, Pauli M, Broekaert I, Classen M, Posovszky C, Schmidt-Choudhury A; im Namen und Auftrag der AGs CEDATA und AG Ernahrung und Diatetik/Ernahrungsmedizin der GPGE. [Crohn's Disease Exclusion Diet - an alternative to exlusive enteral nutritional therapy in children and adolescents with Crohn's disease? Statement of the GPGE working groups CEDATA and Nutrition/Nutrition Medicine]. Z Gastroenterol. 2020 Sep;58(9):890-894. doi: 10.1055/a-1199-6751. Epub 2020 Sep 18. German. PMID 32947634
- [Background] Buderus S, Scholz D, Behrens R, Classen M, De Laffolie J, Keller KM, Zimmer KP, Koletzko S; CEDATA-GPGE Study Group. Inflammatory bowel disease in pediatric patients: Characteristics of newly diagnosed patients from the CEDATA-GPGE Registry. Dtsch Arztebl Int. 2015 Feb 20;112(8):121-7. doi: 10.3238/arztebl.2015.0121. PMID 25759978
- [Background] Bruckner A, Werkstetter KJ, de Laffolie J, Wendt C, Prell C, Weidenhausen T, Zimmer KP, Koletzko S; CEDATA-GPGE study group. Incidence and Risk Factors for Perianal Disease in Pediatric Crohn Disease Patients Followed in CEDATA-GPGE Registry. J Pediatr Gastroenterol Nutr. 2018 Jan;66(1):73-78. doi: 10.1097/MPG.0000000000001649. PMID 28604511
- [Background] Leiz M, Knorr M, Moon K, Tischler L, Sohrabi K, Cantez S, Dabritz J, de Laffolie J, van den Berg N; CEDATA GPGE Study Group. How can patient registries facilitate guideline-based healthcare? A retrospective analysis of the CEDATA-GPGE registry for pediatric inflammatory bowel disease. BMC Health Serv Res. 2023 Jun 17;23(1):648. doi: 10.1186/s12913-023-09639-6. PMID 37330476
- [Background] Schneider N, Sohrabi K, Schneider H, Zimmer KP, Fischer P, de Laffolie J; CEDATA-GPGE Study Group. Machine Learning Classification of Inflammatory Bowel Disease in Children Based on a Large Real-World Pediatric Cohort CEDATA-GPGE(R) Registry. Front Med (Lausanne). 2021 May 24;8:666190. doi: 10.3389/fmed.2021.666190. eCollection 2021. PMID 34109197
- [Background] Peters S, Cantez S, De Laffolie J; CEDATA Study Group. Implementation of exclusive enteral nutrition in pediatric patients with Crohn's disease-results of a survey of CEDATA-GPGE reporting centers. Mol Cell Pediatr. 2022 Apr 5;9(1):6. doi: 10.1186/s40348-022-00139-x. PMID 35381916
- [Background] Classen M, de Laffolie J, Classen M, Schnell A, Sohrabi K, Hoerning A. Significant advantages for first line treatment with TNF-alpha inhibitors in pediatric patients with inflammatory bowel disease - Data from the multicenter CEDATA-GPGE registry study. Front Pediatr. 2022 Jul 19;10:903677. doi: 10.3389/fped.2022.903677. eCollection 2022. PMID 36304532
- [Background] Laffolie J, Zimmer KP, Sohrabi K, Hauer AC. Early Immune Suppression in Children and Adolescents With Crohn's Disease-Data From the CEDATA GPGE Registry. Dtsch Arztebl Int. 2021 Jun 18;118(24):421-422. doi: 10.3238/arztebl.m2021.0214. No abstract available. PMID 34369371
- [Background] De Laffolie J, Ballauff A, Wirth S, Blueml C, Rommel FR, Classen M, Laass M, Lang T, Hauer AC; CEDATA-GPGE Study Group. Occurrence of Thromboembolism in Paediatric Patients With Inflammatory Bowel Disease: Data From the CEDATA-GPGE Registry. Front Pediatr. 2022 Jun 3;10:883183. doi: 10.3389/fped.2022.883183. eCollection 2022. PMID 35722497
- [Background] Elonen L, Wolfle L, de Laffolie J, Posovszky C; CEDATA-GPGE-Study-Group. Isolated Crohn's Colitis: Is Localization Crucial? Characteristics of Pediatric Patients From the CEDATA-GPGE Registry. Front Pediatr. 2022 May 31;10:875938. doi: 10.3389/fped.2022.875938. eCollection 2022. PMID 35712614
- [Background] Leiz M, Knorr M, Moon K, Tischler L, de Laffolie J, van den Berg N. Diagnostic delay in children with inflammatory bowel disease in the German-Austrian patient registry CEDATA-GPGE 2014-2018. Sci Rep. 2022 Dec 7;12(1):21162. doi: 10.1038/s41598-022-25487-6. PMID 36477258
- [Background] Klamt J, de Laffolie J, Wirthgen E, Stricker S, Dabritz J; CEDATA-GPGE study group. Predicting complications in pediatric Crohn's disease patients followed in CEDATA-GPGE registry. Front Pediatr. 2023 Feb 15;11:1043067. doi: 10.3389/fped.2023.1043067. eCollection 2023. PMID 36873644
- See also: Login Page — https://cedata-v2.fb11.uni-giessen.de/login
- See also: Description and Newsletter (german) — https://www.gpge.eu/forschungespghan